CLINICAL TRIAL: NCT07233876
Title: A Prospective, Multi-Center, Single-Arm Study for the Evaluation of the DuOCor 2 Ventricular Assist SysteM In Patients With AdvaNced BIventriCulAr HearT FailurE
Brief Title: DuoCor 2 DOMINATE Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Core Medical Technology CO.,LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COREMED_EU_DuoCor
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Advanced Heart Failure
Keywords: Mechanical Circulatory Support; Biventricular Heart Failure; Biventricular Assist Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DuoCor VAS (Experimental): The DuoCor Ventricular Assist System (DuoCor VAS) to be used on patients with advanced biventricular heart failure
  Interventions: Device: DuoCor Ventricular Assist System

INTERVENTIONS:
Device: DuoCor Ventricular Assist System — Implantation of the DuoCor Ventricular Assist System for mechanical circulatory support.

SUMMARY:
Advanced heart failure is a life-threatening condition characterized by the inability of one or both ventricles to maintain adequate blood circulation. In such cases, medical treatments often prove ineffective, necessitating advanced treatment. Heart transplantation is the standard treatment for these patients, but it is severely limited by the shortage of donor hearts. As a result, mechanical circulatory support (MCS) devices are often employed. However, the most common form, the left ventricular assist device (LVAD), is only suitable for patients with isolated left ventricular dysfunction. This leaves a significant treatment gap for patients with biventricular failure. For this population, current options, such as total artificial hearts (TAHs) and biventricular assist devices (BiVADs), are associated with significant challenges, including high rates of adverse events and suboptimal long-term outcomes.

The DuoCor Ventricular Assist System (VAS) is a next-generation MCS device specifically developed to address this need by providing simultaneous biventricular support. It incorporates two compact, good hemocompatible blood pumps designed for implantation in both the left and right heart, controlled via a single driveline and external controller. It aims to reduce surgical complexity, improve patient mobility, and minimize complications such as thrombosis and infection.

The primary objective of this study is to evaluate the safety and efficacy of the DuoCor VAS as a treatment for advanced biventricular heart failure.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years and ≤ 75 years
* 2. Patient is inotrope dependent, OR has a Cardiac Index (CI) < 2.2 L/min/m2, while not on inotropes
* 3. Patient has left heart failure with at least one of the following criteria:
* Left ventricular ejection fiction (LVEF) ≤ 30%;
* Pulmonary capillary wedge pressure (PCWP) > 15mmHg.
* 4. Patient has severe, irreversible biventricular heart failure and is eligible for biventricular mechanical circulatory support based on the ISHLT guideline. This includes at least two of the following hemodynamic and/or echocardiographic measurements:
* Right ventricular ejection fraction (RVEF)≤ 30%;
* Right ventricular stroke work index (RVSWI)≤ 0.25 mmHg*L/m2;
* Tricuspid annular plane systolic excursion (TAPSE)≤ 14 mm;
* Right ventricular (RV) to left ventricular (LV) end-diastolic diameter ratio> 0.72;
* Central venous pressure (CVP)> 15 mmHg;
* CVP to PCWP ratio> 0.63;
* Tricuspid insufficiency grade 2-4;
* Pulmonary artery pressure index (PAPi)< 2;
* 5. Patient or its legal representative has signed the informed consent, has full understanding of procedures and the study, and is committed to following study requirements.

Exclusion Criteria:

* 1. Known intolerance to anticoagulant or antiplatelet therapies.
* 2. Etiology of heart failure due to restrictive or constrictive physiology (e.g., hypertrophic cardiomyopathy, cardiac amyloidosis /senile or other infiltrative heart disease).
* 3. Coagulopathy defined by platelets < 100k/µl or INR ≥ 1.5 not due to anticoagulant therapy.
* 4. Technical obstacles which pose an inordinately high surgical risk, in the judgment of the investigator.
* 5. Presence of temporary mechanical circulatory support such as Impella (all types) or IABP with a duration greater than 21 days.
* 6. Presence of ECMO with a duration greater than 10 days.
* 7. Patient is implanted with durable mechanical circulatory support (LVAD or RVAD) and has refused to switch to the study device.
* 8. Patient experienced cerebrovascular accident (CVA) within 3 months of eligibility evaluation.
* 9. Presence of any one of the following risk factors for indications of severe end organ dysfunction or failure:
* Total bilirubin > 3.0 mg/dL or cirrhosis confirmed by imaging or positive biopsy;
* Glomerular filtration rate (GFR) < 30 mL/min/1.73 m2 or renal replacement therapy dependence;
* History of severe chronic obstructive pulmonary disease (COPD) defined by FEV1/FVC < 0.7, or FEV1 < 50% predicted.
* Significant peripheral vascular disease (PVD) accompanied by rest pain or extremity ulceration;
* 10. Fixed pulmonary hypertension with a most recent PVR ≥ 8 Wood units.
* 11. Severe systemic light-chain amyloidosis.
* 12. Blood stream infection within seven days. Positive blood cultures reflective of contaminants (e.g., Staphylococcus epidermidis) will not be considered an exclusion.
* 13. Sepsis
* 14. History of confirmed, untreated abdominal aortic aneurysm (AAA) or thoracic aortic aneurysm (TAA) > 5 cm in diameter.
* 15. Any condition other than HF that could limit survival to less than 24 months.
* 16. Positive pregnancy test if of childbearing potential.
* 17. Lactating mothers.
* 18. Participation in any other clinical investigation that is likely to confound study results or affect the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Composite of survival at 6 months post-implantation | 6 months
  At 6 months post-implantation, composite of survival to transplant, recovery (defined that the removal/switch off all the pump of the DuoCor VAS due to the cardiac recovery), or survival with the device (whether with one or both pumps).

SECONDARY OUTCOMES:
Function Status as measured by Six Minute Walk Test (6MWT) | Baseline, Month 3, Month 6
  The more meters a patient can walk over baseline indicates improvement in functional status.
Functional status as measured by the New York Heart Association (NYHA) Classification | Baseline, Month 3, Month 6
  NYHA class categorizes patients by the severity of their heart failure symptoms. As the class increases, the degree of symptoms is more severe indicating worse functional status.
Quality of Life as measured by the EuroQoL-5D-5L (EQ-5D-5L) | Baseline, Month 3, Month 6
  The scores from the 5 dimensions are summed for the total score which ranges from 5 to 25 with higher scores indicating more problems and a worse quality of life.
Quality of Life as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ) | Baseline, Month 3, Month 6
  The scores range from 0 to 100. Higher scores indicate better quality of life and fewer heart failure symptoms.
Adverse Events | As they occurred, from Baseline to Month 6
  Frequency and incidence of all anticipated Adverse Event as defined in (INTERMACS Adverse Events Definition Date: 10/11/2021)

CONTACTS AND LOCATIONS:
Overall Officials: Jan D Schmitto, Principal Investigator — Hannover Medical School
Locations (1):
- Medizinische Hochschule Hannover, Hanover, Germany

IPD SHARING:
Plan to Share IPD: Undecided
At this moment the IPD is not yet available for access and will be updated when it is ready.